CLINICAL TRIAL: NCT03064841
Title: Clinical Characteristics, Anti-hyperglycaemic Treatment Pattern and Target Attainment of Type 2 Diabetes Mellitus Patients in Older Population With or Without Albuminuria in China: A Nationwide Cross-sectional Study
Brief Title: Clinical Characteristics, Anti-hyperglycaemic Treatment Pattern and Target Attainment of Type 2 Diabetes Mellitus Patients in Older Population With or Without Albuminuria in China
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1218.174
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Outpatient with confirmed T2DM: subjects with confirmed T2DM
  Interventions: Drug: No Treatment

INTERVENTIONS:
Drug: No Treatment — No treatment

SUMMARY:
This is a multi-centre, cross-sectional, non-interventional study assessing blood glucose target attainment, anti-hyperglycaemic treatment pattern and the clinical characteristics in older outpatients with Type 2 Diabetes Mellitus (T2DM) in hospitals of China. This study is designed to collect information of older T2DM patients in a real life setting

ELIGIBILITY:
Inclusion criteria

* Patient should fully know and understand the content of consent form, and the patient is willing and able to sign an informed consent form
* Outpatient with confirmed T2DM (According to the American Diabetes Association criteria 2015 [R16-1532])
* Age≥60 years

Exclusion criteria

* Patients with type 1 diabetes mellitus or secondary DM
* Patients who are participating in any other clinical study, including any questionnaire-based study, any interventional study (including diet/counselling based intervention), or any clinical study in which any medications (including Chinese herbal medications) are administered

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 1500 patients will be recruited with Type 2 Diabetes Mellitus consecutively from departments of endocrinology from at least 30 hospitals of China.
Sampling Method: Non-Probability Sample
Enrollment: 1537 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (18):
- China (18):
  - Peking University Shougang Hospital, Beijing
  - Beijing Hospital, Beijing
  - Beijing Pinggu Hospital, Beijing
  - China Meitan General Hospital, Beijing
  - First Hospital of Jilin University, Changchun
  - Chinese Traditional Medicine Hospital of Sichuna Provinc, Chengdu
  - West China Hospital, Chengdu
  - First Affiliated Hospital of Dalian Medical University, Dalian
  - Forth Clinical Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Nanjing First Hospital, Nanjing
  - Integrated Chinese and Western Medicine Hospital, Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - The affiliated hospital of medicalcollege qingdao university, Qingdao
  - Shengjing Hospital of China Medical University, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited into the study in the order of their clinical visits scheduled. First 7 consented and suitable patients were recruited for each site on each day, or fewer if without enough patients. One study visit was planned for each patient.The data was collected for this study from 09th March, 2017 to 30th December, 2017.
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be included in the study if any of specific entry criteria was violated.
Groups:
- Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM): Outpatients with confirmed type 2 diabetes mellitus (T2DM), whose treatments patterns included only diet control and exercise; oral antidiabetic drug (OAD)-mono therapy; OAD-combined therapy; insulin only; OAD and insulin both.
Period: Overall Study
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Started | 1537
Completed | 1520
Not Completed | 17
Not completed — Inclusion/exclusion criteria violation | 4
Not completed — No glycated haemoglobinA1c measurement | 11
Not completed — Screen failure | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set - Eligible (FAS - E):
  The FAS - E includes all eligible patients regarding to inclusion and exclusion criteria with an glycated haemoglobin A1c (HbA1c) measurement.
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.7 (5.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 819
  Male | 701
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Attained Blood Glucose Control Target Defined as Glycated Haemoglobin A1c (HbA1c)<7%, According to 2015 American Diabetes Association (ADA) and 2013 Chinese Diabetes Society (CDS) Guidelines.
Description: The percentage of patients attaining blood glucose control target defined as HbA1c<7%, according to 2015 American Diabetes Association (ADA) and 2013 Chinese Diabetes Society (CDS) guidelines.
Time Frame: At study visit (one day)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
Percentage of patients | 43.4

2. Secondary Outcome: Renal Function Level of Patients Measured by Albuminuria
Description: The renal function level of patients was measured by albuminuria into following categories - normal, micro-albuminuria, macro-albuminuria and missing data.
  Albuminuria was measured using either as a random spot urine sample, a 24-h urine sample, or a timed urine sample. Normal was defined as < 30 mg/g, <30 mg/24h, and < 20 μg/min with the random spot urine sample, the 24-h urine sample, and the timed urine sample, respectively. Micro-albuminuria was defined as 30 - 300 mg/g, 30 - 300 mg/24h, and 20 - 200 μg/min with the random spot urine sample, the 24-h urine sample, and the timed urine sample, respectively. Macro-albuminuria was defined as >300 mg/g, >300 mg/24h, and >200 μg/min with the random spot urine sample, the 24-h urine sample, and the timed urine sample, respectively.
Time Frame: At study visit (one day)
Population: FAS - E
Measure: Number; unit: Percentage of patients
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
Percentage of patients
  Normal | 63.8
  Micro-albuminuria | 27.6
  Macro-albuminuria | 7.1
  Missing | 1.5

3. Secondary Outcome: Renal Function Level of Patients Measured by Estimated Glomerular Filtration Rate (eGFR)
Description: The renal function level of patients was measured by estimated glomerular filtration rate (eGFR).
Time Frame: At study visit (one day)
Population: FAS - E
Measure: Mean (Standard Deviation); unit: milliLitre/minute/1.73 meter ^ 2
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
milliLitre/minute/1.73 meter ^ 2 | 85.019 (18.204)

4. Secondary Outcome: Renal Function Level of Patients Measured by Chronic Kidney Disease (CKD) Stage
Description: The renal function level of patients was measured by CKD into following categories - eGFR ≥ 60 milliLitre/minute/1.73 meter ^ 2 (mL/min/1.73m^2), eGFR < 60 mL/min/1.73m^2 and missing data.
Time Frame: At study visit (one day)
Population: FAS - E
Measure: Number; unit: Percentage of patients
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
Percentage of patients
  eGFR >=60 mL/min/1.73m^2 | 51.1
  eGFR < 60 mL/min/1.73m^2 | 5.4
  Missing eGFR data | 43.6

5. Secondary Outcome: Treatment Regimens for T2DM That Patient Are Currently Taking
Description: The treatment regimens for T2DM that patient are currently taking.
Time Frame: At study visit (one day)
Population: FAS - E
Measure: Number; unit: Percentage of patients
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
Percentage of patients
  No treatment | 2.6
  Only diet control and exercise | 7.5
  Oral antidiabetic drug (OAD) - Mono therapy | 16.8
  OAD - Combined therapy | 28.7
  Insulin only | 15.5
  OAD and Insulin | 28.3
  Missing | 0.6

6. Secondary Outcome: Percentage of Patients Macro-vascular and Micro-vascular Diabetic Complications
Description: The percentage of patients macro-vascular and micro-vascular diabetic complications.
Time Frame: At study visit (one day)
Population: FAS - E
Measure: Number; unit: Percentage of patients
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
Percentage of patients
  Cardiovascular disease | 14.9
  Cerebrovascular disease | 11.2
  Peripheral vascular disease | 8.8
  Kidney disease | 8.6
  Retinopathy | 14.4
  Neuropathy | 13.6

7. Secondary Outcome: Percentage of Patients With Hypoglycaemic Occurrence
Description: The percentage of patients with hypoglycaemic occurrence.
Time Frame: At study visit (one day)
Population: FAS - E
Measure: Number; unit: Percentage of patients
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
Percentage of patients | 28.0

8. Secondary Outcome: Percentage of Patients With Hypoglycaemia Leading to Therapy Change
Description: The percentage of patients with hypoglycaemia leading to therapy change.
Time Frame: At study visit (one day)
Population: FAS - E
Measure: Number; unit: Percentage of patients
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
Percentage of patients | 7.2

9. Secondary Outcome: Percentage of Patients With Anti-hypertension Therapy Usage
Description: The percentage of patients with anti-hypertension therapy usage.
Time Frame: At study visit (one day)
Population: FAS - E
Measure: Number; unit: Percentage of patients
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
Percentage of patients | 49.0

10. Secondary Outcome: Percentage of Patients With Lipid Lowering Therapy Usage
Description: The percentage of patients with lipid lowering therapy usage.
Time Frame: At study visit (one day)
Population: FAS - E
Measure: Number; unit: Percentage of patients
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
Percentage of patients | 29.2

11. Secondary Outcome: Percentage of Patients With Anti-platelet Therapy Usage
Description: The percentage of patients with anti-platelet therapy usage.
Time Frame: At study visit (one day)
Population: FAS - E
Measure: Number; unit: Percentage of patients
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
Percentage of patients | 30.1

12. Secondary Outcome: Follow up Duration of Type 2 Diabetes Related Risk Factors in Clinical Practice
Description: The follow up duration of type 2 diabetes related risk factors was summarized using the situation of lab test including serum creatinine, uric acid, high density lipoprotein cholesterol, low density lipoprotein cholesterol, triglyceride and total cholesterol.
Time Frame: At study visit (one day)
Population: FAS - E
Measure: Number; unit: Percentage of patients
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
Number analyzed (Participants) | 1520
Percentage of patients
  Follow-up duration - within 3 months | 33.6
  Follow-up duration - within 3 to 6 months | 16.1
  Follow-up duration - within 6 to 12 months | 17.3
  Follow-up duration - More than 12 months | 27.8
  Missing follow-up duration | 5.3

ADVERSE EVENTS:
Time Frame: From signing the informed consent until completed the visit that day i.e., up to 24hrs.
Description: Due to the non-interventional character of this study and since there was no requirement for the patients to use a kind of BI drug, only all adverse drug reactions (ADRs), all adverse events (AEs) with fatal outcome and spontaneously mentioned safety events were to be collected as required.
Arm/Group | Outpatients With Confirmed Type 2 Diabetes Mellitus (T2DM)
All-Cause Mortality (participants affected / at risk) | 0/1520
Serious Adverse Events (participants affected / at risk) | 0/1520
Other Adverse Events (participants affected / at risk) | 0/1520

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT03064841/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT03064841/SAP_001.pdf